CLINICAL TRIAL: NCT00431912
Title: A Multicenter Open Label Phase II Study of to Assess the Efficacy and Safety of APO866 in the Treatment of Patients With Refractory or Relapsed Cutaneous T-cell Lymphoma
Brief Title: A Study of APO866 for the Treatment of Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP3001
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: cutaneous T-cell lymphoma; mycosis fungoides; Sézary syndrome; APO866; phase II study
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — N-(4-(1-benzoylpiperidin-4-yl)butyl)-3-(pyridin-3-yl)acrylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm, trinomial 2-stage design (Experimental)
  Interventions: Drug: APO866

INTERVENTIONS:
Drug: APO866 — APO866 is administered as 0.126 mg/m²/hr for 4 consecutive days (96 hours), every 3 weeks for a total of 3 cycles

SUMMARY:
This phase II study is designed to determine the efficacy and safety of APO866 for the treatment of patients with advanced forms of cutaneous T-cell lymphoma (CTCL). APO866 has shown to induce growth inhibition in cultures of human CTCL cells as well as in animal models with subcutaneously implanted human CTCL tumors. APO866 was considered to be safe and well-tolerated in a phase I study that treated 24 patients with advanced cancer. APO866 is administered by intravenous infusion continuously for 96 hours and that is repeated every 4 weeks. Patients will receive 3 cycles of treatment and the primary efficacy endpoint will be assessed at Week 16. patients will be followed up for 12 months

DETAILED DESCRIPTION:
CTCL is the most frequent occurring cutaneous non-Hodgkin lymphoma characterized by an indolent and protracted course of patches, plaques and tumors. It is highly symptomatic, debilitating, disfiguring and impacting on the patient's quality of life. The treatment strategy for CTCL is based on the exact diagnosis including the stage of disease and aims to preserve cellular immune function, while achieving an anti-tumor effect. Given the nature of the disease and the cumulative and additive toxicities of treatments used, the intensity and duration of long-term therapy is limited.

APO866 is novel drug that induces cell death by specifically inhibiting the biosynthesis of NAD+ from niacinamide, which is essential for the cellular metabolism, protein modification (e.g. PARP mediated DNA repair, sirtuins (histone deacetylation)) and Calcium dependent messenger synthesis. APO866 is not subject to the commonly known mechanisms of MDR. Its activity is cell cycle independent. APO866 exerted high anti-tumor activity on a broad range of different tumor cells derived from both human solid cancers and leukemias in vitro and on large number of human xenografts in nude mice and rats in vivo. Hematologic cancer cells were highly sensitive to APO866. Lymphocytes are the most sensitive normal cells to APO866 resulting to lymphocytopenia and reticulocytopenia in rats, monkeys and cancer patients. Furthermore, APO866 may have anti-angiogenic properties as shown in vivo and in patients.

APO866 has shown to induce, at low nM level, growth inhibition of human Myla CTCL cells as well as in human subcutaneous xenografts of Myla CTCL in Balb-C nude mice.

APO866 was investigated in 24 patients with advanced cancers in a phase I study aiming to determine the DLT and MTD. Treatment was well tolerated and safe. The unique DLT was thrombocytopenia. At dose levels higher than 0.036 mg/m2/hr CTC grade III lymphocytopenia, thought not be clinically relevant, preceded all other toxicities. The recommended dose for phase II studies of APO866 is 0.126 mg/m2/hr administered by civ infusion for 4 consecutive days (MTD). This dose was selected because of its safety profile, and the translational observation that Css of APO866 at MTD was similar or higher as compared to the concentrations at which efficacy was established in vitro and in vivo.

No objective tumor response was observed. However, 4 patients had stable disease for at least 3 months: prostate cancer (4 months), melanoma (5 months), sarcomatoid mesothelioma (3 months) and oropharyngeal cancer (5 months). In addition, lesion size reductions were observed in the melanoma patient (80% size reduction and stable size of other lesions) at an APO866 dose level of 0.072 mg/m2/hr, and in the mesothelioma patient (moderate size reductions of pleural lesions) at 0.108 mg/m2/hr.

Treatment with APO866 was safe and well tolerated. The anti-tumor effect of APO866, in particular on hematological cancer cells in vitro and ex vivo, and its lymphocytopenic effect in patients support the rationale to conduct an open phase II study of APO866 in patients with refractory or relapsed CTCL qualifying for systemic chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of CTCL including mycosis fungoides and Sézary syndrome
* Stage Ib to IVb disease (AJCC TNM staging, see Appendix B)
* Relapsed or refractory disease or intolerant to ≥ 2 prior systemic therapy. PUVA, topical nitrogen mustard, spot or total skin electron beam therapy or other radiotherapy, oral retinoids, immunotherapy (e.g. interferon-α, denileukin difitox, alemtuzumab) or mono- or poly-chemotherapy regimen will be considered systemic therapy.
* ECOG Performance Status < 2 (see Appendix C)
* Age > 18 years, of either sex
* Female patients with childbearing potential must be using a hormonal contraceptive, intra uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study. Women of childbearing potential must have a negative serum or urinary hCG pregnancy test
* Male patients, who are not surgically sterile, must use a condom with spermicide for the duration of the study
* Have given written informed consent, prior to any study related procedure not part of the patient's normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Have participated in any other investigational study or received an experimental therapeutic procedure considered to interfere with the study in the 2 months preceding SD1
* Have had PUVA, topical nitrogen mustard, spot or total skin electron beam therapy, oral retinoids, or any, immunotherapy (e.g. interferon-α, denileukin difitox, alemtuzumab) or chemotherapy regimen within 2 weeks of SD1. Patients must have recovered from all acute toxicities.
* Evidence of CNS lymphoma
* Use of prohibited medication due to CYP3A4 metabolism of APO866, as specified in Section 6.6.2. concomitant use of these drugs will not be allowed during the study.
* Uncontrolled medical conditions, requiring surgical or pharmacological treatment (exceptions must be approved by the Study Director).
* Serious concomitant disease (e.g. significant cardiac disease) are not eligible
* Primary or acquired thrombocytopenia
* Inadequate bone marrow reserve: WBC < 3.5x10^9/L, neutrophils < 1.0x10^9/L, thrombocytes < 100x10^9/L, Hb < 8.5 g/dL or coagulation abnormalities
* Inadequate liver function: total bilirubin > 1.5 x upper limit of normal values (ULN), AST, ALT, or alkaline phosphatase > 2.5 x ULN
* Have inadequate renal function, defined by serum creatinine > 250 μmol/L
* Retinopathy, history of retinal laser surgery, or an ERG < 50% of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The proportion of eligible patients with refractory or relapsed CTCL whom have a complete response or partial response on cutaneous lesions (Tumor Burden Index) and extra-cutaneous disease. | Week 16

SECONDARY OUTCOMES:
Safety and tolerability, time to response, duration of overall response, duration of stable disease and time to treatment failure. | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, MD PhD, Principal Investigator — Department of Dermatology, University Hospital of Zürich, Gloriastrasse 31, 8091 Zürich, Switzerland; René Goedkoop, MD, Study Director — Apoxis SA, 18-20 Avenue de Sévelin, 1004 Lausanne, Switzerland
Locations (5):
- Department of Dermatology, Medical University Graz, Graz, Austria
- France (2):
  - Deapartment of Dermatology, Créteil
  - department of Dermatologie, Hotel Dieu, Nantes
- University Clinic for Dermatology, Medical Faculty of Mannheim of the Heidelberg University, Mannheim, Germany
- Department of Dermatology, University Hospital of Zürich, Zurich, Switzerland